CLINICAL TRIAL: NCT04129632
Title: Evaluation of Institutional Job Demands-Resources and a Novel Mindfulness Tool on Burnout Intensity in a Cross-sectional Cohort of Colorado Health Care Practitioners
Brief Title: Evaluation of Institutional Resources and a Novel Mindfulness Tool on Burnout Intensity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkview Medical Center (Other)
Responsible Party: Principal Investigator, Doug Duffee, Internal Medicine Residency Faculty Attending Physician, Parkview Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PIRB67
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Burnout, Professional
Keywords: burnout; wellness; mindfulness; physician burnout
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cross sectional study design with intra cohort voluntary intervention participation
Masking Description: No demographic linking to survey participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IEPF intervention (Other): Survey respondent voluntary decides to do a 4 weeks mindfulness intervention
  Interventions: Behavioral: IEPF Wellness Tool

INTERVENTIONS:
Behavioral: IEPF Wellness Tool — A daily 5 minute mindfulness exercise over 28 days
  Other Names: Insights and Exercises in Personal Forgiveness from Psalm 19

SUMMARY:
: The problem of physician burnout has been well documented. As health care providers (HCP) encounter the demands and resources of a rapidly changing health care system, navigate their place and performance within it, deal with the demands of an internet informed patient populace and balance daily work load with family life, stressors arise. These stressors can contribute to burnout and this burnout has both interpersonal and health care system wide effects. Studies have shown that HCP burnout has personal physiologic consequences and predicts external objective associations with health care acquired infection rates, medical errors, medical litigation, patient satisfaction, job satisfaction, health care system costs, alcohol abuse and suicidal ideation, among others. As our population ages and its medical co-morbidities and system demands increase, the premature curtailing, cessation or turnover of an HCP's clinical practice due to emotional exhaustion is a concerning trend. While studies have shown that HCP's are no more prone to burnout then other professionals, a growing body of literature has shown that an intentional focus on institutional processes that nurture clinician well-being through multiple modalities is both important and effective. Additionally, insights into the role that forgiveness plays in personal well-being prompts our presentation of a novel mindfulness tool that focuses on improving clinician well-being through self-help exercises in meditation and forgiveness. In light of recent studies that have cautioned against the tendency to dichotomize and/or pathologize peoples' responses to their work environment, we will use the JD-R (Job demands-resources model) and the CBI (Copenhagen burnout inventory) to quantify these processes and responses. These factors have prompted us to present a unique study design a) to evaluate the wellness process affecters inside the culture of a regional health care center and b) to evaluate the effectiveness of a personal mindfulness intervention which aims at spectrum based burnout quantification and facilitated self-help, with an eye on both for institution wide application.

DETAILED DESCRIPTION:
Title: Evaluation of Institutional Job Demands-Resources and a Novel Mindfulness Tool on Burnout intensity in a Cross-Sectional Cohort of Colorado Health Care Practitioners Author: Doug Duffee MD, Mdiv, FACP, Attending Physician Parkview Internal Medicine Residency Program, Pueblo Colorado 2019 Intro: The problem of physician burnout has been well documented. As health care providers (HCP) encounter the demands and resources of a rapidly changing health care system, navigate their place and performance within it, deal with the demands of an internet informed patient populace and balance daily work load with family life, stressors arise. These stressors can contribute to burnout and this burnout has both interpersonal and health care system wide effects. Studies have shown that HCP burnout has personal physiologic consequences and predicts external objective associations with health care acquired infection rates, medical errors, medical litigation, patient satisfaction, job satisfaction, health care system costs, alcohol abuse and suicidal ideation, among others. As our population ages and its medical co-morbidities and system demands increase, the premature curtailing, cessation or turnover of an HCP's clinical practice due to emotional exhaustion is a concerning trend. While studies have shown that HCP's are no more prone to burnout then other professionals, a growing body of literature has shown that an intentional focus on institutional processes that nurture clinician well-being through multiple modalities is both important and effective. Additionally, insights into the role that forgiveness plays in personal well-being prompts our presentation of a novel mindfulness tool that focuses on improving clinician well-being through self-help exercises in meditation and forgiveness. In light of recent studies that have cautioned against the tendency to dichotomize and/or pathologize peoples' responses to their work environment, we will use the JD-R (Job demands-resources model) and the CBI (Copenhagen burnout inventory) to quantify these processes and responses. These factors have prompted us to present a unique study design a) to evaluate the wellness process affecters inside the culture of a regional health care center and b) to evaluate the effectiveness of a personal mindfulness intervention which aims at spectrum based burnout quantification and facilitated self-help, with an eye on both for institution wide application.

Aims and Objectives: Using the Health Care Provider Wellness Assessment as quantified through the revised Job Demands-Resources Model (JD-R), the Copenhagen Burnout Inventory (CBI) (20)and a novel mindfulness tool called "Psalm 19: Insights and Exercises in Personal Forgiveness", we propose to 1) Identify unique institutional job demands-resources whose presence-absence contribute to HCP strain and subsequent health impairment and 2) Assess the ability of said novel mindfulness tool as a personal job resource component to positively affect well-being and subsequent job motivation amongst a cohort of Colorado health care providers at a regional medical center. As beneficial process effectors are identified (more/better/culturally focused resources, less/better efficiency demands) , multi-factorial interventions on wellness outcomes can subsequently be studied and implemented.

Methods:

Diagram Current Environment Wellness Process Wellness Outcomes

* Health impairment process Job Demands + >Strain/burnout + >Health Problems l- /- l- \- l- Job Resources + >Well-being/engagement +>Performance
* Motivational process

  1. Design: Single blinded cohort controlled Cross-sectional survey research design using the JD-R, CBI and Wellness Tool to determine associations and affects on HCP burnout

     •identify cross-sectional intervention with survey cohort AND survey only control cohort>>>survey (with or without intervention) >>>analyze data
  2. Population: Colorado health care clinicians (DO, MD, PA, NP, RN, PharmD and MA) at a single regional health care system (PMC) anonymously and voluntarily responding to the Parkview Medical Center Health Care Provider Wellness Assessment
  3. Ethics: Blinded and voluntary participation

Survey:

Parkview Medical Center Health Care Provider Wellness Assessment

1. Parkview Medical Center Process Effectors (from JD-R revised): "on a scale of 1-5 (never/almost never, seldom, sometimes, often, always), rate your interaction with the following:"

   I. Job Demands:
   1. Centralization
   2. Cognitive demands
   3. Complexity
   4. Computer problems
   5. Demanding contact with patients
   6. Downsizing
   7. Emotional demands
   8. Emotional dissonance
   9. Interpersonal conflict
   10. Job insecurity
   11. Negative spillover from family to work
   12. Harassment by patients
   13. Performance demands
   14. Problems planning
   15. Pupil's misbehavior
   16. Qualitative workload
   17. Reorganization
   18. Remuneration
   19. Responsibility
   20. Risks and hazards
   21. Role ambiguity
   22. Role conflict
   23. Sexual harassment
   24. Time pressure
   25. Unfavorable shift and work schedule
   26. Unfavorable work conditions aa. Work pressure bb.Work-home conflict cc.Work overload

   II. Job Resources:

   a. Job based i. Advancement ii. Appreciation iii. Autonomy iv. Craftsmanship v. Financial rewards vi. Goal clarity vii. Information viii. Innovative climate ix. Job challenge x. Knowledge xi. Leadership xii. Opportunities for professional development xiii. Participation in decision making xiv. Performance feedback xv. Positive spillover from family to work xvi. Professional pride xvii. Procedural fairness xviii. Positive patient contacts xix. Quality of the relationship with the supervisor xx. Safety climate xxi. Safety routine violations xxii. Social climate xxiii. Social support from colleagues xxiv. Social support from supervisor xxv. Skill utilization xxvi. Strategic planning xxvii. Supervisory coaching xxviii. Task variety xxix. Team cohesion xxx. Team harmony xxxi. Trust in management b. Personal based i. Emotional and mental competencies ii. Extraversion iii. Hope iv. Intrinsic motivation v. Low neuroticisim vi. Need satisfaction (autonomy, belongingness, competence) vii. Optimism viii. Organization-based self esteem ix. Regulatory focus (prevention and promotion focus x. Resilience xi. Self-efficacy xii. Value orientation (intrinsic and extrinsic values) III. Measurement Outcomes, Negative (for future study, once process effectors are identified and intervened upon)
   1. Absenteeism (self-report and company registered)
   2. Accidents and injuries
   3. Adverse events
   4. Depression
   5. Determination to continue
   6. Unsafe behaviors
   7. Negative work-home interference
   8. Physical ill-health
   9. Psychsomatic health complaints
   10. Psychological strain (General Health Questionairre, GHQ)
   11. Turnover intention IV. Measurement Outcomes, Positive (for future study, once process effectors are identified and intervened upon)

   <!-- -->

   1. Extra-role performance (self or other rated)
   2. Innovativeness
   3. In-role performance (self or other rated)
   4. Life satisfaction
   5. Organizational commitment
   6. Perceived health
   7. Positive work-home interference
   8. Service quality
   9. Team sales performance
   10. Workability
   11. Happiness
2. Copenhagen Burnout Inventory: "on a scale of 1-5 (never/almost never, seldom, sometimes, often, always), rate your interaction with the following:" a. Personal burnout i. How often do you fell tired? ii. How often are you physically exhausted? iii. How often are you emotionally exhausted? iv. How often do you think: "I can't take it anymore"? v. How often do you feel worn out? vi. How often do you feel weak and susceptible to illness? b. Work-related burnout i. Is your work emotionally exhausting? ii. Do you feel burnt out because of your work? iii. Does your work frustrate you? iv. Do you feel worn out at the end of the working day? v. Are you exhausted in the morning at the thought of another day at work? vi. Do you feel that every working hour is tiring for you? vii. Do you have enough energy for family and friends during leisure time? (reverse the scoring: 1-5 is (always, often, sometimes, seldom, never/almost never) c. Client-related burnout i. Do you find it hard to work with clients? ii. Do you find it frustrating to work with clients? iii. Does it drain your energy to work with clients? iv. Do you feel that you give more than you get back when you work with clients? v. Are you tired of working with clients? vi. Do you sometimes wonder how long you will be able to continue working with clients?

ELIGIBILITY:
Inclusion Criteria:

* DO's, MD's, MA's, NP's, PA's, RN's, PharmD's

Exclusion Criteria:

* any one not in the above professional categories

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Copenhagen Burnout Inventory score | 6 months
  A numerical quantification of burnout in health care providers with and without intervention. 19 questions, 1-5 scale, 19-95 total score, higher is worse/more burnout

CONTACTS AND LOCATIONS:
Overall Officials: Doug Duffee, MD, Principal Investigator — Parkview Medical Center
Locations (1):
- Parkview Medical Center, Pueblo, Colorado, United States

REFERENCES:
- [Background] Yaribeygi H, Panahi Y, Sahraei H, Johnston TP, Sahebkar A. The impact of stress on body function: A review. EXCLI J. 2017 Jul 21;16:1057-1072. doi: 10.17179/excli2017-480. eCollection 2017. PMID 28900385
- [Background] Shanafelt TD, Noseworthy JH. Executive Leadership and Physician Well-being: Nine Organizational Strategies to Promote Engagement and Reduce Burnout. Mayo Clin Proc. 2017 Jan;92(1):129-146. doi: 10.1016/j.mayocp.2016.10.004. Epub 2016 Nov 18. PMID 27871627
- [Background] Rotenstein LS, Torre M, Ramos MA, Rosales RC, Guille C, Sen S, Mata DA. Prevalence of Burnout Among Physicians: A Systematic Review. JAMA. 2018 Sep 18;320(11):1131-1150. doi: 10.1001/jama.2018.12777. PMID 30326495
- [Background] Dyrbye et al., Burnout Among Health Care Professionals, A Call to Explore and Address This Under recognized Threat to Safe, High-Quality Care. NAM Perspectives. Discussion Paper, National Academy of Medicine.
- [Background] Henry JP. Biological basis of the stress response. Integr Physiol Behav Sci. 1992 Jan-Mar;27(1):66-83. doi: 10.1007/BF02691093. PMID 1576090
- [Background] McEwen BS. Neurobiological and Systemic Effects of Chronic Stress. Chronic Stress (Thousand Oaks). 2017 Jan-Dec;1:2470547017692328. doi: 10.1177/2470547017692328. Epub 2017 Apr 10. PMID 28856337
- [Background] McEwen BS. Protective and damaging effects of stress mediators. N Engl J Med. 1998 Jan 15;338(3):171-9. doi: 10.1056/NEJM199801153380307. No abstract available. PMID 9428819
- [Background] Health, US report, 2016, CDC.
- [Background] Silver MP, Hamilton AD, Biswas A, Warrick NI. A systematic review of physician retirement planning. Hum Resour Health. 2016 Nov 15;14(1):67. doi: 10.1186/s12960-016-0166-z. PMID 27846852
- [Background] Julkunen J, Salonen R, Kaplan GA, Chesney MA, Salonen JT. Hostility and the progression of carotid atherosclerosis. Psychosom Med. 1994 Nov-Dec;56(6):519-25. doi: 10.1097/00006842-199411000-00007. PMID 7871107
- [Background] Cavanagh K, Strauss C, Forder L, Jones F. Can mindfulness and acceptance be learnt by self-help?: a systematic review and meta-analysis of mindfulness and acceptance-based self-help interventions. Clin Psychol Rev. 2014 Mar;34(2):118-29. doi: 10.1016/j.cpr.2014.01.001. Epub 2014 Jan 10. PMID 24487343
- [Background] Harris, Alex HS., et al, Forgiveness, Unforgiveness, Health and Disease from Handbook of Forgiveness 2005, Routledge, Everett L. Worthington, ed.
- [Background] Thoresen, CE., et al, Effects of Forgiveness Intervention on perceived stress, state and trait anger and self-reported health. Paper presented at annual meeting for society of behavioral health, Seattle WA, 2001.
- [Background] Waltman, MA., The psychological and physiological effects of forgiveness education in male patients with coronary artery disease. Dissertation Abstracts International: Section B: The Sciences and Engineering; 63(8-B), 3971.
- [Background] Witvleit, C., forgiveness and Health: Review and reflections on a matter of faith, feelings and physiology, Journal of Psychology and Theology, 29, 212-224.
- [Background] Witvleit, C., et al., Please forgive me: Transgressors' emotions and physiology during imagery of seeking forgiveness and victim responses. Journal of Psychology and Christianity, 21, 219-233.
- [Background] vanOyen Witvliet C, Ludwig TE, Vander Laan KL. Granting forgiveness or harboring grudges: implications for emotion, physiology, and health. Psychol Sci. 2001 Mar;12(2):117-23. doi: 10.1111/1467-9280.00320. PMID 11340919
- [Background] Worthington EL Jr, Witvliet CV, Pietrini P, Miller AJ. Forgiveness, health, and well-being: a review of evidence for emotional versus decisional forgiveness, dispositional forgivingness, and reduced unforgiveness. J Behav Med. 2007 Aug;30(4):291-302. doi: 10.1007/s10865-007-9105-8. Epub 2007 Apr 24. PMID 17453329
- [Background] Lupano Perugini ML, de la Iglesia G, Castro Solano A, Keyes CL. The Mental Health Continuum-Short Form (MHC-SF) in the Argentinean Context: Confirmatory Factor Analysis and Measurement Invariance. Eur J Psychol. 2017 Mar 3;13(1):93-108. doi: 10.5964/ejop.v13i1.1163. eCollection 2017 Mar. PMID 28344677
- [Background] The Copenhagen Burnout Inventory: A new tool for the assessment of burnout, Work and Stress 19(3): 192-207, July-September 2005
- [Background] Wohl, MMJA et al., Looking Within: Measuring State Self-Forgiveness and Its relationship to Psychological Well-Being. Canadian Journal of Behavioral Science 2008, Vol 40(1): 1-10.
- [Background] Bakker, A B et al., Using the jobs demands-resources model to predict burnout and performance. 2004 Human Resource Management, 43, 83-104.